CLINICAL TRIAL: NCT06587204
Title: Understanding Decentralized Trial Engagement and Clinical Impediments Through Digital Efforts (UDECIDE) Among Unrepresented Groups With Poor Cardiovascular and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Azizi Seixas, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20240230
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (Other): Participants in this group will be receiving the standard of care for up to 3 months.
  Interventions: Other: Control Group
- Decentralized Group (Experimental): Participants in this group will be receiving the decentralized intervention for up to 3 months.
  Interventions: Behavioral: Decentralized Group
- Digital Literacy Navigation Group (Experimental): Participants in this group will be receiving the Digital Literacy Navigation intervention for up to 3 months.
  Interventions: Behavioral: Decentralized Group; Behavioral: Digital Literacy Navigation Group
- Social Care Navigation Group (Experimental): Participants in this group will be receiving the Social Care Navigation intervention for up to 3 months.
  Interventions: Behavioral: Decentralized Group; Behavioral: Digital Literacy Navigation Group; Behavioral: Social Care Navigation Group

INTERVENTIONS:
Other: Control Group — Participants will receive standard of care.
  Arms: Control Group
Behavioral: Decentralized Group — Participants will receive a one time digital lifestyle management program that will be used for the rest of the intervention. The Digital lifestyle management program is a virtual application that manages nutrition, exercise, and sleep. Participants will be using the application at least 1 hour each day.
  Arms: Decentralized Group; Digital Literacy Navigation Group; Social Care Navigation Group
Behavioral: Digital Literacy Navigation Group — Participants will receive a one time digital literacy training virtual learning digital health education for the rest of the intervention . The digital literacy training is a digital health education program that will be given 1 hour a day for 3 weeks.
  Arms: Digital Literacy Navigation Group; Social Care Navigation Group
Behavioral: Social Care Navigation Group — Participants will receive a one time social care navigation application that will be used for the rest of the intervention. The Social Care Navigation application is a digital application that provides social care resources in the community to participants. The application is used 1 hour a day, each day.
  Arms: Social Care Navigation Group

SUMMARY:
The objective of the UDECIDE study is to demonstrate adherence to decentralized clinical trials among underrepresented groups with cardiometabolic conditions .

ELIGIBILITY:
Inclusion Criteria:

* History of pre-diabetes/diabetes and/or pre-hypertension/hypertension
* History of Cardiometabolic risk factors including the following: hypertension, Coronary Artery Disease (CAD), heart attack, heart failure, stroke, atherosclerosis, arrhythmias, Peripheral Artery Disease (PAD), type 2 diabetes, metabolic syndrome, obesity, dyslipidemia, insulin resistance, or elevated cholesterol.
* Identify as Black or non-White Hispanic
* Own a smart phone

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants adhering to the intervention | 3 months
  Will be measured in percentage
Percentage of participants retained in the intervention | 3 months
  Will be measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Azizi Seixas, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No